CLINICAL TRIAL: NCT01342978
Title: Human Papillomavirus (HPV) Oral Transmission Study in Partners Over Time
Acronym: HOTSPOT
Status: Completed | Type: Observational
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: Icahn School of Medicine at Mount Sinai (Other); Oregon Health and Science University (Other); Dana-Farber Cancer Institute (Other); Johns Hopkins University (Other)
Responsible Party: Principal Investigator, Gypsyamber D'Souza, Associate Professor, Johns Hopkins Bloomberg School of Public Health
Other Study IDs: HOTSPOT
Record Dates: First submitted 2011-03-07; First posted 2011-04-27 (Estimated); Last update posted 2017-03-03 (Actual); Status verified 2017-02

CONDITIONS: Oropharyngeal Cancer; Human Papillomavirus
Keywords: HPV; HNSCC
MeSH Terms: conditions — Oropharyngeal Neoplasms; Squamous Cell Carcinoma of Head and Neck

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples With DNA — Serum, oral rinse/saliva and some tumor samples
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (3):
- oropharyngeal cancer case: 208 oropharyngeal cancer cases were enrolled
- partner or spouse of case: 110 partners of patients with oropharyngeal cancer were enrolled
- control: A convenience group of 106 non-cancer controls were enrolled at some study sites at cancer screening events

SUMMARY:
This research is being done to understand more about a sexually transmitted virus called Human papillomavirus (HPV) in people with oropharyngeal cancer and their partners.

DETAILED DESCRIPTION:
This study evaluates oral HPV infection and risk factors in people with head and neck cancer and their partners or spouses. The study focuses on oropharyngeal cancer patients and includes patients with HPV-associated and HPV-unassociated disease. A comparison group of people without cancer (controls) are also being enrolled. Couples are followed longitudinally and there is a repository of study samples. It is hoped that this research will help us understand risk factors for oral HPV infection, persistence and transmission as well as researching biomarkers for HPV-associated oral cancer and survival.

The study is led by Dr Amber D'Souza (Johns Hopkins) and laboratory testing for the study is performed in the laboratory of study co-investigator Dr Maura Gillison (Ohio University). The study biorepository is led by Dr karen Anderson (Arizona State). Participants are being enrolled at four sites across the United States including: Mt Sinai (site PI Dr Marshall Posner), Johns Hopkins (site PI Dr Sara Pai), Dana Farber Cancer Institute (site PI Dr Robert Haddad) and Oregon Health and Science University (site PI Dr Neil Gross).

ELIGIBILITY:
Inclusion Criteria:

* 18 years or older and incident oropharyngeal cancer

Exclusion Criteria:

* Presence of medical or psychiatric condition affecting ability to give voluntary, informed consent
* Cancer patients with a history of organ transplant, autoimmune disorder treated with steroids or immunosuppressive drug, lymphoma, leukemia or bone marrow transplant are also ineligible (partners with these conditions are eligible)

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: cohort of cancer patients with matched enrollment of spouses and non-cancer controls
Sampling Method: Non-Probability Sample
Enrollment: 242 (Actual)
Dates: Start 2009-10; Primary Completion 2014-12 (Actual); Study Completion 2017-01 (Actual)

PRIMARY OUTCOMES:
HPV DNA detection in oral rinse sample | baseline
  Detection of 17 types of HPV DNA in exfoliated oral cells of cases and partners collected using an oral rinse and gargle

CONTACTS AND LOCATIONS:
Overall Officials: Gypsyamber D'Souza, PhD, Principal Investigator — Johns Hopkins Bloomberg School of Public Health
Locations (4):
- United States (4):
  - Johns Hopkins Hospital, Baltimore, Maryland
  - Dana Farber Cancer Institute, Boston, Massachusetts
  - Mt Sinai School of Medicine, New York, New York
  - Oregon Health & Science University, Portland, Oregon

REFERENCES:
- [Result] Anderson KS, Wong J, D'Souza G, Riemer AB, Lorch J, Haddad R, Pai SI, Longtine J, McClean M, LaBaer J, Kelsey KT, Posner M. Serum antibodies to the HPV16 proteome as biomarkers for head and neck cancer. Br J Cancer. 2011 Jun 7;104(12):1896-905. doi: 10.1038/bjc.2011.171. PMID 21654689
- [Result] D'Souza G, Gross ND, Pai SI, Haddad R, Anderson KS, Rajan S, Gerber J, Gillison ML, Posner MR. Oral human papillomavirus (HPV) infection in HPV-positive patients with oropharyngeal cancer and their partners. J Clin Oncol. 2014 Aug 10;32(23):2408-15. doi: 10.1200/JCO.2014.55.1341. Epub 2014 Apr 28. PMID 24778397